CLINICAL TRIAL: NCT03995784
Title: Phase 2b Study to Evaluate the Pharmacokinetics, Pharmacodynamics, Efficacy and Safety of a Subcutaneous Prophylaxis Treatment Regimen of CB2679d, in Adult Subjects With Hemophilia B
Brief Title: Study of Next-Generation Recombinant Factor IX Variant in Adult Subjects With Hemophilia B
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalyst Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DLZ-201
Record Dates: First submitted 2019-06-19; First posted 2019-06-24 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Dose (Experimental): Coagulation Factor IX variant, 50 IU/kg by intravenous route
  Interventions: Biological: Coagulation Factor IX variant
- Subcutaneous Dosing (Experimental): Coagulation Factor IX variant, 100 IU/kg by subcutaneous route
  Interventions: Biological: Coagulation Factor IX variant

INTERVENTIONS:
Biological: Coagulation Factor IX variant — Single intravenous injection of CB2679d/Dalcinonacog alfa
  Arms: Intravenous Dose
Biological: Coagulation Factor IX variant — Daily subcutaneous injections of CB2679d/Dalcinonacog alfa for 28 days
  Arms: Subcutaneous Dosing

SUMMARY:
Phase 2b, single-center, open-label study designed to evaluate the pharmacokinetics, pharmacodynamics, efficacy and safety of subcutaneous (SC) prophylaxis treatment regimens with CB2679d in 6 adult, male subjects with severe congenital hemophilia B.

DETAILED DESCRIPTION:
Single-center, open-label Phase 2b study will evaluate the PK, PD, efficacy and safety parameters of SC prophylaxis treatment regimens with CB2679d in adult subjects with hemophilia B. The study will enroll and dose subcutaneously, a total of 6 adult male subjects with severe congenital hemophilia B.

During the Treatment Period, the subject will receive an IV dose of 50 IU/kg followed 35 ± 5 minutes later by a SC dose of 100 IU/kg. Daily SC doses of 100 IU/kg will be administered until Day 28 (28 total SC doses). On Day 1, PK, PD, and safety assessments will be done at pre-IV dose and repeated 35 (± 5) minutes later prior to the SC dose. Subsequent PK, PD and safety assessments will be performed pre-dose on days 2, 3, 7, 14, 21 and 28.

During the Washout Period, PK, PD, and safety assessments will be done on Days 29, 30, 31, 32 and 33. Daily FIX activity levels will be measured, unless FIX activity level is known to be < 5%, as measured by local laboratory.

An End of Study visit will occur 30 days (± 2 days) after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of severe (<2%) congenital hemophilia B.
* Male, age 18 or older.
* Agreement to use highly effective birth control throughout the study.
* Affirmation of informed consent with signature confirmation before any trial-related activities.
* Stated willingness to comply with all study procedures and availability for the duration of the study.

Exclusion Criteria:

* History or a family history of FIX inhibitors.
* Positive antibody to FIX detected by central laboratory at screening.
* Previous participation in and subsequent treatment in a clinical trial within the previous 30 days or 3-half-lives, whichever is longer, or absence of clinical effect.
* Have a coagulation disorder other than congenital hemophilia B.
* Factor IX gene mutation 128G>A.
* Significant contraindication to participation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Levy, MD, PhD, MMM, Study Director — Catalyst Biosciences
Locations (1):
- Haemophilia Comprehensive Care Centre, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: No
This is a single-center, open label study so the investigator will have full access to all study subject data.

REFERENCES:
- [Derived] Faraj A, Le Moan N, Gorina E, Blouse GE, Knudsen T, Simonsson USH. Model-Informed Support of Dose Selection for Prophylactic Treatment with Dalcinonacog Alfa in Adult and Paediatric Hemophilia B Patients. Adv Ther. 2023 Sep;40(9):3739-3750. doi: 10.1007/s12325-023-02570-6. Epub 2023 Jun 21. PMID 37341915

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 subjects were screened in the study, but 4 subjects failed screening due to inclusion/exclusion criteria not met and 1 subject was screened, but withdrew consent before receiving any study medication. These 5 subjects were considered not enrolled into the Treatment Period, and the remaining 6 were considered enrolled into the Treatment Period. Of those 6 enrolled into the Treatment Period, 5 subjects completed the study. The 6 subjects enrolled comprise the Overall Subjects/Population.
Groups:
- Overall Subjects: Subjects were dosed with a single intravenous injection dose of 50 IU/kg coagulation Factor IX variant (CB2679d/Dalcinonacog alfa) and then daily subcutaneous doses of 100 IU/kg coagulation Factor IX variant (CB2679d/Dalcinonacog alfa) for 28 days
Period: Overall Study
Arm/Group | Overall Subjects
Started | 6
Completed | 5
Not Completed | 1
Not completed — One subject discontinued on Day 7 due to injection site reactions after Day 1, 2, and 3 doses | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Subjects: All subjects in the Safety Population received study treatment
Arm/Group | Overall Subjects
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved FIX Level ≥12%
Description: Subjects who achieved a FIX activity level ≥12% during the treatment period in the PK Population
Time Frame: Days 7, 14, 21, 28, 29
Population: PK population. One subject not included in the PK population discontinued the study on Day 7 and had an activity level >12%
Measure: Count of Participants; unit: Participants
Groups:
- Overall Subjects: All subjects in the PK population
Arm/Group | Overall Subjects
Number analyzed (Participants) | 5
Participants
  Day 7 | 3
  Day 14 | 4
  Day 21 | 4
  Day 28 | 4
  Day 29 | 5

2. Secondary Outcome: FIX Activity Levels (Actual and Change From Baseline) in All Subjects
Description: FIX Activity Levels measured by percent activity.
  Baseline was defined as the lowest assessment before the first administration of study drug. Maximum change from baseline was calculated as the maximum of the changes from baseline over all visits during treatment period. FIX activity level below the limit of quantification (BLQ) were set to zero. In case of retest, the average of the different test results were considered for the summary analyses.
  1 subject received a higher IV dose than allowed per protocol (150 IU/kg) at Day 1 thus this subject's values at Day 1 (SC Dose), Day 2, & Day 3 were excluded from this analysis & the total number of participants was lowered by 1 at these timepoints. Additionally, mean (standard deviation) for the maximum change from baseline in the FIX activity level (%) during SC dosing was calculated by excluding actual values at Day 1 IV dose, Day 1 SC dose, Day 2 & Day 3 for all 6 subjects.
Time Frame: Screening, Day 1 (IV Pre-dose, SC Dose), Day 2, 3, 7, 14, 21, 28, 29, 30, 31, 32, 33, and End of Study. End of Study is the average of each subject's last recorded assessment (between Days 29 to 33).
Population: PK Population. 1 subject received a higher IV dose than allowed per protocol (150 IU/kg) at Day 1 thus this subject's values at Day 1 (SC Dose), Day 2, & Day 3 were excluded from this analysis & the total number of participants was lowered by 1 at these timepoints. Additionally, mean (standard deviation) for the maximum change from baseline in the FIX activity level (%) during SC dosing was calculated by excluding actual values at Day 1 IV dose, Day 1 SC dose, Day 2 & Day 3 for all 6 subjects.
Measure: Mean (Standard Deviation); unit: % (percent) activity
Groups:
- Actual Value (%): Actual Values of FIX activity levels during study
- Change From Baseline (%): Change from Baseline in values of FIX activity levels during study
Arm/Group | Actual Value (%) | Change From Baseline (%)
Number analyzed (Participants) | 5 | 5
% (percent) activity
  Screening: number analyzed (Participants) | 5 | 0
  Screening | 0.24 (0.5367) |
  Day 1, IV Predose: number analyzed (Participants) | 5 | 0
  Day 1, IV Predose | 11.54 (20.3775) |
  Day 1, SC Dose: number analyzed (Participants) | 4 | 4
  Day 1, SC Dose | 25.538 (9.2245) | 25.238 (8.7156)
  Day 2: number analyzed (Participants) | 4 | 4
  Day 2 | 15.05 (4.7177) | 14.75 (4.1589)
  Day 3: number analyzed (Participants) | 4 | 4
  Day 3 | 13.8 (2.7362) | 13.5 (2.5153)
  Day 7 | 13.64 (4.7141) | 13.4 (4.7974)
  Day 14 | 18.66 (7.7986) | 18.42 (7.5301)
  Day 21 | 18.74 (6.5328) | 18.5 (6.1895)
  Day 28 | 19.92 (6.6571) | 19.68 (6.3622)
  Day 29 | 19.44 (4.385) | 19.2 (4.1905)
  Day 30 | 14.92 (3.4354) | 14.68 (3.2653)
  Day 31 | 12.06 (1.8119) | 11.82 (1.4721)
  Day 32 | 8.763 (2.7348) | 8.463 (2.3085)
  Day 33 | 8.288 (1.7148) | 7.988 (1.1707)
  End of Study | 0.32 (0.7155) | 0.08 (0.1789)
  SC Maximum change from baseline during SC dosing: number analyzed (Participants) | 0 | 5
  SC Maximum change from baseline during SC dosing |  | 21.183 (4.4723)

3. Secondary Outcome: Pharmacokinetic (PK) Analysis - AUC
Description: Summary of Pharmacokinetic Parameters - AUC Infinity Observation and AUC to Last Non-zero Concentration
Time Frame: From date of first dose of CB2679d until date of first occurrence of clinical event, assessed up to treatment Day 28. PK sampling was conducted on Day 1 (IV pre-dose -5 min, SC 30 min post IV dose, hour 7 +/- 1 hour) and Day 2 (hour 24 +/- 1 hour).
Population: PK Population
Measure: Mean (Standard Deviation); unit: IU/dL*day
Groups:
- Area Under the Curve (AUC): Observations of mean PK parameters
Arm/Group | Area Under the Curve (AUC)
Number analyzed (Participants) | 5
IU/dL*day
  AUC Infinity Observation | 126.0306 (26.80093)
  AUC to Last Non-zero Concentration | 75.415 (17.22908)

4. Secondary Outcome: PK Analysis - Clearance
Description: Summary of PK Parameters - Clearance
Time Frame: as for outcome 3
Population: PK Population
Measure: Mean (Standard Deviation); unit: dL/day/kg
Groups:
- Value: Observations of mean PK parameters
Arm/Group | Value
Number analyzed (Participants) | 5
dL/day/kg | 0.8191544 (0.15349536)

5. Secondary Outcome: PK Analysis - Maximum Concentration During SC Dosing
Description: Summary of PK Parameters - Maximum Concentration during SC dosing
Time Frame: as for outcome 3
Population: PK Population
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Value
Number analyzed (Participants) | 5
IU/dL | 20.74 (5.58)

6. Secondary Outcome: PK Analysis - Half-Life and Residence Time
Description: Summary of PK Parameters - Half-Life-1(alpha), Half-Life-1(beta), and Mean Residence Time
Time Frame: as for outcome 3
Population: PK Population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Value
Number analyzed (Participants) | 2
days
  Half-Life-1(alpha) | 5.32395 (3.049964)
  Half-Life-1(beta) | 3.87172 (1.132563)
  Mean Residence Time | 6.1572 (1.609332)

7. Secondary Outcome: PK Analysis - Volume of Distribution at Steady-State Observed
Description: Summary of PK Parameters - Volume of Distribution at Steady-State Observed
Time Frame: as for outcome 3
Population: PK Population
Measure: Mean (Standard Deviation); unit: dL/kg
Arm/Group | Value
Number analyzed (Participants) | 5
dL/kg | 5.00736 (1.542769)

8. Secondary Outcome: Occurrence of Clinical Thrombotic Event
Description: Rate of occurrence of clinical thrombotic event not attributable to another cause
Time Frame: From date of first dose of CB2679d until date of first occurrence of clinical event, assessed up to treatment Day 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Overall Safety Population: All subjects in the Safety Population received study treatment
Arm/Group | Overall Safety Population
Number analyzed (Participants) | 6
Participants | 0

9. Secondary Outcome: Occurrence of an Antibody Response
Description: Rate of occurrence of an antibody response to CB2679d and cross-reactive with wild-type recombinant coagulation FIX
Time Frame: From date of first dose of CB2679d until date of first occurrence of clinical event, assessed up to treatment Day 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Safety Population
Number analyzed (Participants) | 6
Participants
  Confirmed Antidrug Antibody (ADA) to DalcA | 2
  Neutralizing antibody to DalcA | 0

10. Secondary Outcome: Thrombogenicity Assessment - Fibrinogen
Description: Evaluation of the levels of thrombogenicity markers of a subcutaneous regimen of CB2679d
Time Frame: as for outcome 2
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Actual Value: Actual Values during study
- Change From Baseline: Change from Baseline in values during study
Arm/Group | Actual Value | Change From Baseline
Number analyzed (Participants) | 5 | 5
mg/dL
  Fibrinogen - Screening: number analyzed (Participants) | 5 | 0
  Fibrinogen - Screening | 300.4 (64.77) |
  Fibrinogen - Day 1, IV Pre-dose: number analyzed (Participants) | 5 | 0
  Fibrinogen - Day 1, IV Pre-dose | 305.6 (73.53) |
  Fibrinogen - Day 1, SC Dose | 326.4 (79.04) | 20.8 (12.50)
  Fibrinogen - Day 2 | 296.2 (72.29) | -9.4 (18.04)
  Fibrinogen - Day 3 | 299.2 (65.98) | -6.4 (33.58)
  Fibrinogen - Day 7 | 285.8 (52.64) | -19.8 (71.92)
  Fibrinogen - Day 14 | 272.2 (42.81) | -33.4 (87.16)
  Fibrinogen - Day 21 | 283.6 (55.68) | -22.0 (78.19)
  Fibrinogen - Day 28 | 314.4 (87.21) | 8.8 (149.17)
  Fibrinogen - Day 29 | 313.2 (73.31) | 7.6 (141.32)
  Fibrinogen - Day 30 | 306.0 (62.38) | 0.4 (127.73)
  Fibrinogen - Day 31 | 313.8 (76.40) | 8.2 (138.79)
  Fibrinogen - Day 32: number analyzed (Participants) | 4 | 4
  Fibrinogen - Day 32 | 300.8 (114.93) | 22.8 (107.82)
  Fibrinogen - Day 33: number analyzed (Participants) | 4 | 4
  Fibrinogen - Day 33 | 342.8 (68.75) | 64.8 (87.93)
  Fibrinogen - End of Study | 285.2 (30.60) | -20.4 (101.45)
  Fibrinogen - Maximum change from baseline during dosing: number analyzed (Participants) | 0 | 5
  Fibrinogen - Maximum change from baseline during dosing |  | -10.4 (103.83)

11. Secondary Outcome: Thrombogenicity Assessment - D-Dimer
Description: Evaluation of the levels of thrombogenicity markers of a subcutaneous regimen of CB2679d
Time Frame: as for outcome 2
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Actual Value | Change From Baseline
Number analyzed (Participants) | 5 | 5
ug/L
  D-Dimer - Screening: number analyzed (Participants) | 5 | 0
  D-Dimer - Screening | 169.6 (155.63) |
  D-Dimer - Day 1, IV Pre-dose: number analyzed (Participants) | 5 | 0
  D-Dimer - Day 1, IV Pre-dose | 218.6 (153.78) |
  D-Dimer - Day 1, SC Dose | 209.6 (183.77) | -9.0 (58.71)
  D-Dimer - Day 2 | 654.6 (426.46) | 436.0 (427.86)
  D-Dimer - Day 3 | 680.6 (405.82) | 462.0 (378.00)
  D-Dimer - Day 7 | 761.0 (550.10) | 542.4 (572.80)
  D-Dimer - Day 14 | 969.4 (993.15) | 750.8 (1053.87)
  D-Dimer - Day 21 | 772.6 (999.62) | 554.0 (1069.36)
  D-Dimer - Day 28 | 590.8 (311.30) | 372.2 (410.31)
  D-Dimer - Day 29 | 675.6 (845.00) | 457.0 (920.85)
  D-Dimer - Day 30 | 313.4 (275.43) | 94.8 (343.02)
  D-Dimer - Day 31 | 293.8 (242.76) | 75.2 (314.13)
  D-Dimer - Day 32: number analyzed (Participants) | 4 | 4
  D-Dimer - Day 32 | 364.5 (371.95) | 143.5 (433.31)
  D-Dimer - Day 33: number analyzed (Participants) | 4 | 4
  D-Dimer - Day 33 | 390.5 (323.83) | 169.5 (404.25)
  D-Dimer - End of Study | 212.8 (177.26) | -5.8 (242.12)
  D-Dimer - Maximum change from baseline during dosing: number analyzed (Participants) | 0 | 5
  D-Dimer - Maximum change from baseline during dosing |  | 1088.0 (921.99)

12. Secondary Outcome: Thrombogenicity Assessment - Prothrombin Fragments 1 + 2
Description: Evaluation of the levels of thrombogenicity markers of a subcutaneous regimen of CB2679d
Time Frame: as for outcome 2
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Actual Value | Change From Baseline
Number analyzed (Participants) | 5 | 5
pmol/L
  Prothrombin Fragments 1 + 2 - Screening: number analyzed (Participants) | 5 | 0
  Prothrombin Fragments 1 + 2 - Screening | 151.2 (55.63) |
  Prothrombin Fragments 1 + 2 - Day 1, IV Pre-dose: number analyzed (Participants) | 5 | 0
  Prothrombin Fragments 1 + 2 - Day 1, IV Pre-dose | 187.8 (126.73) |
  Prothrombin Fragments 1 + 2 - Day 1, SC Dose | 195.2 (141.90) | 7.4 (58.11)
  Prothrombin Fragments 1 + 2 - Day 2 | 171.4 (75.79) | -16.4 (93.75)
  Prothrombin Fragments 1 + 2 - Day 3 | 158.8 (63.08) | -29.0 (88.88)
  Prothrombin Fragments 1 + 2 - Day 7 | 203.2 (110.30) | 15.4 (129.60)
  Prothrombin Fragments 1 + 2 - Day 14 | 192.8 (99.38) | 5.0 (130.70)
  Prothrombin Fragments 1 + 2 - Day 21 | 126.6 (39.63) | -61.2 (127.21)
  Prothrombin Fragments 1 + 2 - Day 28 | 151.2 (51.44) | -36.6 (98.34)
  Prothrombin Fragments 1 + 2 - Day 29 | 120.4 (36.86) | -67.4 (138.05)
  Prothrombin Fragments 1 + 2 - Day 30 | 117.2 (33.11) | -70.6 (118.47)
  Prothrombin Fragments 1 + 2 - Day 31 | 122.0 (40.38) | -65.8 (111.81)
  Prothrombin Fragments 1 + 2 - Day 32: number analyzed (Participants) | 4 | 4
  Prothrombin Fragments 1 + 2 - Day 32 | 112.5 (27.06) | -83.5 (148.20)
  Prothrombin Fragments 1 + 2 - Day 33: number analyzed (Participants) | 4 | 4
  Prothrombin Fragments 1 + 2 - Day 33 | 124.5 (33.51) | -71.5 (122.25)
  Prothrombin Fragments 1 + 2 - End of Study | 115.6 (27.76) | -72.2 (143.95)
  Prothrombin Fragments 1 + 2 - Maximum change from baseline during dosing: number analyzed (Participants) | 0 | 5
  Prothrombin Fragments 1 + 2 - Maximum change from baseline during dosing |  | -16.8 (178.49)

13. Secondary Outcome: Thrombogenicity Assessment - Thrombin/Antithrombin
Description: Evaluation of the levels of thrombogenicity markers of a subcutaneous regimen of CB2679d
Time Frame: as for outcome 2
Population: Pharmacodynamic Population
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | Actual Value | Change From Baseline
Number analyzed (Participants) | 5 | 5
ug/L
  Thrombin/Antithrombin - Screening: number analyzed (Participants) | 5 | 0
  Thrombin/Antithrombin - Screening | 9.34 (13.518) |
  Thrombin/Antithrombin - Day 1, IV Pre-dose: number analyzed (Participants) | 4 | 0
  Thrombin/Antithrombin - Day 1, IV Pre-dose | 1.93 (1.130) |
  Thrombin/Antithrombin - Day 1, SC Dose | 4.42 (2.724) | 2.14 (1.692)
  Thrombin/Antithrombin - Day 2 | 3.86 (1.053) | 1.58 (1.134)
  Thrombin/Antithrombin - Day 3 | 3.86 (0.808) | 1.58 (0.993)
  Thrombin/Antithrombin - Day 7 | 5.08 (2.745) | 2.80 (2.677)
  Thrombin/Antithrombin - Day 14 | 6.72 (4.017) | 4.44 (3.686)
  Thrombin/Antithrombin - Day 21 | 4.08 (1.279) | 1.80 (1.873)
  Thrombin/Antithrombin - Day 28 | 6.38 (4.581) | 4.10 (3.707)
  Thrombin/Antithrombin - Day 29 | 3.36 (0.841) | 1.08 (1.561)
  Thrombin/Antithrombin - Day 30 | 3.24 (0.684) | 0.96 (0.733)
  Thrombin/Antithrombin - Day 31 | 8.52 (13.498) | 6.24 (12.939)
  Thrombin/Antithrombin - Day 32: number analyzed (Participants) | 4 | 4
  Thrombin/Antithrombin - Day 32 | 3.88 (2.244) | 1.63 (1.941)
  Thrombin/Antithrombin - Day 33: number analyzed (Participants) | 4 | 4
  Thrombin/Antithrombin - Day 33 | 4.05 (2.447) | 1.80 (2.008)
  Thrombin/Antithrombin - End of Study | 3.62 (1.547) | 1.34 (2.726)
  Thrombin/Antithrombin - Maximum change from baseline during dosing: number analyzed (Participants) | 0 | 5
  Thrombin/Antithrombin - Maximum change from baseline during dosing |  | 5.44 (2.581)

ADVERSE EVENTS:
Time Frame: TEAEs were defined as AEs that occurred on or after the first dose of study medication or worsened after the first dose of study drug in this study but not later than the date of last dose (+30 days).
Arm/Group | Overall Subjects
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Subjects (N=6)
Injection Site Reaction (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT03995784/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/84/NCT03995784/SAP_001.pdf